CLINICAL TRIAL: NCT01809847
Title: Ofatumumab Induction and Maintenance in Elderly Patients With Poor Risk CLL in the Context of Allogeneic Transplantation(CLL-X4 Trial)
Brief Title: Ofatumumab Induction and Maintenance in Elderly Patients With Poor Risk CLL in the Context of Allogeneic Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Dresden (Other); University Hospital Ulm (Other); University Hospital Schleswig-Holstein (Other); University Hospital of Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUD-CLL-X4-054; 2012-001947-31 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2013-03-13 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Lymphatic Leukemia
Keywords: CLL; Chronic Lymphatic Leukemia; Leukemia; HLA; Histocompatibility; HCT; hematopoietic stem cell transplantation; Ofatumumab; CD20
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): First dose of 300 mg Ofatumumab followed by seven weekly infusions of 2000 mg. Dexamethasone will be given orally at doses of 40 mg on days 1-4 in weeks 1, 3, 5, and 7. Maintenance therapy consists of 6 monthly infusions of 1000 mg ofatumumab.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — Study treatment comprises eight weeks of induction therapy with ofatumumab in combination with high-dose dexamethasone. The first dose of ofatumumab is 300 mg followed by seven infusions of 2000 mg ofatumumab. Dexamethasone will be given orally at doses of 40 mg on days 1-4 in weeks 1, 3, 5, and 7. Patients who achieved a CR, PR shall proceed to maintenance therapy. Maintenance therapy consists of 6 monthly infusions of 1000 mg ofatumumab.
  An HLA-matched sibling donor or HLA-matched unrelated donor can be identified for approximately 70% of patients. Donor search will be completed within six weeks for 95% of the patients. Patients with a donor will proceed to allogeneic HCT as soon as possible prior to, or during maintenance therapy.
  Other Names: Arzerra; Anti-CD20 antibody

SUMMARY:
To study the safety and efficacy of anti-CD20 blockade with ofatumumab in the context of allogeneic HCT in CLL

DETAILED DESCRIPTION:
The goal of the study is to investigate the safety and efficacy of a consequent anti-CD20 therapy with the antibody ofatumumab in the context of allogeneic HCT. Allogeneic HCT itself is not a study intervention and is triggered by the availability of an HLA-compatible stem cell donor. The study is divided into an induction part and a maintenance part. During induction where the antibody is combined with high dose dexamethasone, the main goal is to reduce the tumor load prior to allogeneic HCT. Patients who achieved disease control (CR, PR and SD) by the antibody proceed to maintenance therapy with the antibody. Patients with progressive disease go off study. The idea behind maintenance therapy is that ofatumumab may contribute to tumor control early after allogeneic stem cell transplantation while T-cell based graft-versus leukemia effects are still not fully established. External tumor control could lower the pressure to taper immunosuppressive drugs early after transplantation and could thereby indirectly contribute to better GVHD-prophylaxis. Furthermore, anti-CD20 antibodies have proven activity in the treatment of chronic GVHD. In summary, the concept of a consequent CD20 blockade in the context of allogeneic transplantation could result in better leukemic control and better GVHD prophylaxis, which is a highly attractive goal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL according to WHO criteria (Hallek 2008) confirmed by flow cytometry of peripheral blood or bone marrow
* Age > 55 years
* Poor-risk disease according to the EBMT CLL Transplant Consensus

  * Non-response or early relapse (within 12 months) after purine analogue-containing therapy
  * Relapse (within 24 months) after purine analogue combination therapy or treatment of similar efficacy (ie, autologous stem cell transplantation)
  * p53 deletion/mutation (del 17p-) requiring treatment
* Measurable disease in the peripheral blood defined by a minimum clonal lymphocyte count of 0.5 GPT/L at the time of study inclusion
* Medically fit patients eligible for allogeneic HCT
* Informed consent for related and unrelated donor search and the goal to perform allogeneic HCT
* Sexually mature males must agree to use adequate and medically accepted method of contraception throughout the study if their sexual partners are woman of child bearing potential (WOCBP) WOCBP must be using an adequate and medically accepted method of contraception to avoid pregnancy throughout the study and for at least 3 months after the study.
* WOCBP includes any female that has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >12 consecutive months); or woman on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level >35mlU/mL.
* WOCBP must have a negative serum or urine pregnancy test prior to the start of the study.

Exclusion Criteria:

* Richter's transformation in current relapse or active disease
* Prior allogeneic HCT
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or participation in any other interventional clinical study
* Non-response to monotherapy with ofatumumab prior to study inclusion
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (left ventricular ejection fraction < 50%)
* Abnormal renal function defined by an estimated GFR < 50 ml/min
* Abnormal lung function tests defined by a DLCO <50%, FEV1%VC <70% despite appropriate treatment
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg or HBcAb
* Positive serology for hepatitis C (HC) defined as a positive test for anti-HCV, confirmed by PCR
* Screening laboratory values:

  * total bilirubin >1.5 times upper normal limit (unless due to AIHA or a known history of Gilbert's disease)
  * ALT or AST >2.5 times upper normal limit
  * Gamma glutamyl transpeptidase (GGT) >2.5 times upper normal limit (unless due to disease involvement of the liver)
* Other past or current hematologic or solid organ malignancy. Subjects who have been free of malignancy for at least 3 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.
* Pregnant or lactating woman
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Response rate after induction therapy | week 9
  efficacy analysis of anti-CD20 blockade with ofatumumab
rate of MRD-negative patients | baseline, week 9, month 14
  rate of MRD-negative patients who did not experience relapse, progression or death within the first 14 months after study enrollment

SECONDARY OUTCOMES:
Rate of allogeneic HCT | month 9
  Rate of patients who reach allogeneic HCT if HLA-matched donor is available
adverse drug reactions grade III/IV | week 1 till week 9; month 4 till month 9; month 12; month 14; until 30 days after last administration of the study medication
Overall, event-, and progression free survival | week 1 till week 9; month 4 till month 9; month 12; month 14; up to 5 years follow-up
relapse incidence | month 4 till month 9; month 12; month 14; up to 5 years follow-up
non-relapse mortality | week 1 till week 9; month 4 till month 9; month 12; month 14; up to 5 years follow-up
Incidences of acute and chronic GVHD | during maintenance therapy; month 12, month 14; up to 5 years follow-up
  provided that allogeneic HCT was conducted

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schetelig, PD Dr. med., Principal Investigator — Universitätsklinikum Carl Gustav Carus, Medizinische Klinik und Poliklinik I, 01307 Dresden
Locations (11):
- Germany (11):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Städtisches Klinikum München Schwabing, München, Bavaria
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder), Brandenburg
  - Deutsche Klinik für Diagnostik, Wiesbaden, Hesse
  - Universitätsmedizin Göttingen, Göttingen, Lower Saxony
  - Klinikum der Universität zu Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Klinikum der Johannes Gutenberg Universität, Mainz, Rhineland-Palatinate
  - Klinikum Chemnitz GmbH, Chemnitz, Saxony
  - Universitätsklinikum Dresden, Dresden, Saxony

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website Study Alliance Leukemia (coordinating study group) — http://www.sal-aml.org